CLINICAL TRIAL: NCT00804583
Title: Genetic Modifiers of CF Liver Disease
Brief Title: Genetic Modifiers of Cystic Fibrosis (CF) Liver Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 01-1421; R01DK066368 (NIH)
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis; Liver Disease
Keywords: Cystic Fibrosis; Liver Disease; Genetic Modifiers
MeSH Terms: conditions — Cystic Fibrosis; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A one time blood draw of 35 mls
Oversight: Data Monitoring Committee: No

SUMMARY:
This study examines "modifier genes" that may play a role in the development of CF liver disease. Modifier genes are genes, other than the CF gene (CFTR), which may directly or indirectly have an affect on how the body responds to the conditions that develop as the result of the defective CFTR gene. Scientists have wondered why some patients with CF develop CF liver disease and why some patients with CF do not. To better understand the problem, this study was designed to examine the genetic makeup of CF patients who are considered to have severe liver disease to see if they can identify any modifier genes. Researchers will study blood samples, pulmonary function tests, and other medical information in hopes that a connection can be made between genetic make-up and how severe the liver disease is. The identification of modifier genes that influence disease severity may ultimately lead to a better understanding of CF liver disease, and may be useful in the development of new treatments.

DETAILED DESCRIPTION:
The clinical heterogeneity in cystic fibrosis (CF) is only partly explained by mutations in the CFTR gene. Most CF patients have evidence of liver dysfunction and focal biliary cirrhosis (fibrosis), and a subset of these patients (5-7%) progresses to severe liver disease (CFLD), as defined by portal hypertension and multilobular cirrhosis. The development of CFLD has no relationship to specific CFTR mutations or other biomarkers, and there is currently no way to identify which CF infants will develop severe liver disease.

The central hypothesis of this proposal is that the development of CFLD reflects the influence of non-CFTR "modifier" alleles (genes). This project is designed to identify associations between non-CFTR genes and CFLD, and test the biological effect of selected alleles on hepatic fibrosis in transgenic murine models. We hypothesize that polymorphisms in multiple genes, each with a conceptual or mechanistic link to liver disease, increase the risk for developing end-stage CF liver disease, and that interactions among these risk factors will define the pathophysiology of this disorder. To achieve our goals, we will study 400 CF patients with well-documented severe liver disease and portal hypertension, and 400 gender and genotype-matched CF patients > age 15 years who have no evidence of CFLD. We propose to identify heritable risk factors for the development of CFLD by evaluation of functional sequence variants within, and single nucleotide polymorphisms associated with, multiple genes associated with CFLD pathogenesis. To test ("validate") the biological effects (impact) of selected genetic alleles on liver fibrosis, we will develop transgenic mice homozygous for DeltaF508 (DF508), who are also expressing an additional candidate gene modifier allele. Better definition of the complex genotypes that increase risk for severe liver disease in CF will allow early identification of CF infants predisposed to develop end-stage liver disease, and thereby allow testing of currently available therapies. Better understanding of the pathobiology of hepatic fibrosis in CF will identify novel targets to prevent (or reduce) the development of CFLD.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with CF, regardless of genotype and age, who have "severe" liver disease with portal hypertension (big spleen, i.e. "splenomegaly" and/or presence of enlarged vessels in the esophagus, i.e. esophageal varices) may be eligible to participate. This would include any person who has been evaluated for a liver transplant, or has already received a liver transplant.

Exclusion Criteria:

* History of Alcohol Abuse
* History of Biliary Atresia
* History of Clinically Significant Hepatitis Infection
* History of Hepatic Vein Thrombosis
* History of Liver Cancer
* History of Portal Vein Thrombosis
* History of Clinically Significant use of total parenteral nutrition (TPN)
* History of Wilson's Disease

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF and liver disease
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2004-03; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
This is not an interventional study | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Wanda K O'Neal, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Mencin A, Seki E, Osawa Y, Kodama Y, De Minicis S, Knowles M, Brenner DA. Alpha-1 antitrypsin Z protein (PiZ) increases hepatic fibrosis in a murine model of cholestasis. Hepatology. 2007 Nov;46(5):1443-52. doi: 10.1002/hep.21832. PMID 17668872
- [Background] Bartlett JR, Friedman KJ, Ling SC, Pace RG, Bell SC, Bourke B, Castaldo G, Castellani C, Cipolli M, Colombo C, Colombo JL, Debray D, Fernandez A, Lacaille F, Macek M Jr, Rowland M, Salvatore F, Taylor CJ, Wainwright C, Wilschanski M, Zemkova D, Hannah WB, Phillips MJ, Corey M, Zielenski J, Dorfman R, Wang Y, Zou F, Silverman LM, Drumm ML, Wright FA, Lange EM, Durie PR, Knowles MR; Gene Modifier Study Group. Genetic modifiers of liver disease in cystic fibrosis. JAMA. 2009 Sep 9;302(10):1076-83. doi: 10.1001/jama.2009.1295. PMID 19738092
- [Background] Friedman, K.J., S.C. Ling, E.M. Lange, M. Macek, Jr., A.J. Handler, R.G. Pace, F. Zou, D.R. Mack, S.C. Bell, G. Castaldo, F. Salvatore, U. Ozcelik, B. Tuemmler, M. Sinaasappel, J.L. Colombo, H. Kayserova, M. Phillips, J. Zielenski, L. Tsui, M.L. Drumm, L.M. Silverman, F.A Wright, P.R Durie, M.R. Knowles, Genetic Modifiers of Severe Liver Disease in Cystic Fibrosis, Pediatr Pulmonol Suppl 28:247:170, 2005.
- [Background] Friedman, K.J., S.C. Ling, E.M. Lange, M. Macek, Jr., A.J. Handler, R.G. Pace, F. Zou, S.C. Bell, G. Castaldo, F. Salvatore, C. Colombo, M.J. Phillips, J. Zielenski, L.C. Tsui, M.L. Drumm, L.M. Silverman, F.A Wright, P.R Durie, M.R. Knowles, Genetic Modifiers of Severe Liver Disease in Cystic Fibrosis, 55th Annual Meeting The American Society of Human Genetics, Salt Lake City, UT, 395:2176/F, 2005.
- [Background] Sun L, Rommens JM, Corvol H, Li W, Li X, Chiang TA, Lin F, Dorfman R, Busson PF, Parekh RV, Zelenika D, Blackman SM, Corey M, Doshi VK, Henderson L, Naughton KM, O'Neal WK, Pace RG, Stonebraker JR, Wood SD, Wright FA, Zielenski J, Clement A, Drumm ML, Boelle PY, Cutting GR, Knowles MR, Durie PR, Strug LJ. Multiple apical plasma membrane constituents are associated with susceptibility to meconium ileus in individuals with cystic fibrosis. Nat Genet. 2012 May;44(5):562-9. doi: 10.1038/ng.2221. PMID 22466613
- [Background] Knowles MR, Drumm M. The influence of genetics on cystic fibrosis phenotypes. Cold Spring Harb Perspect Med. 2012 Dec 1;2(12):a009548. doi: 10.1101/cshperspect.a009548. PMID 23209180
- [Background] Blackman SM, Commander CW, Watson C, Arcara KM, Strug LJ, Stonebraker JR, Wright FA, Rommens JM, Sun L, Pace RG, Norris SA, Durie PR, Drumm ML, Knowles MR, Cutting GR. Genetic modifiers of cystic fibrosis-related diabetes. Diabetes. 2013 Oct;62(10):3627-35. doi: 10.2337/db13-0510. Epub 2013 May 13. PMID 23670970
- [Background] Stonebraker JR, Ooi CY, Pace RG, Corvol H, Knowles MR, Durie PR, Ling SC. Features of Severe Liver Disease With Portal Hypertension in Patients With Cystic Fibrosis. Clin Gastroenterol Hepatol. 2016 Aug;14(8):1207-1215.e3. doi: 10.1016/j.cgh.2016.03.041. Epub 2016 Apr 5. PMID 27062904
- [Background] Polineni D, Piccorelli AV, Hannah WB, Dalrymple SN, Pace RG, Durie PR, Ling SC, Knowles MR, Stonebraker JR. Analysis of a large cohort of cystic fibrosis patients with severe liver disease indicates lung function decline does not significantly differ from that of the general cystic fibrosis population. PLoS One. 2018 Oct 11;13(10):e0205257. doi: 10.1371/journal.pone.0205257. eCollection 2018. PMID 30307979
- [Background] Raraigh KS, Aksit MA, Hetrick K, Pace RG, Ling H, O'Neal W, Blue E, Zhou YH, Bamshad MJ, Blackman SM, Gibson RL, Knowles MR, Cutting GR. Complete CFTR gene sequencing in 5,058 individuals with cystic fibrosis informs variant-specific treatment. J Cyst Fibros. 2022 May;21(3):463-470. doi: 10.1016/j.jcf.2021.10.011. Epub 2021 Nov 12. PMID 34782259
- [Background] Rosenfeld M, Faino AV, Onchiri F, Aksit MA, Blackman SM, Blue EE, Collaco JM, Gordon WW, Pace RG, Raraigh KS, Zhou YH, Cutting GR, Knowles MR, Bamshad MJ, Gibson RL. Comparing encounter-based and annualized chronic pseudomonas infection definitions in cystic fibrosis. J Cyst Fibros. 2022 Jan;21(1):40-44. doi: 10.1016/j.jcf.2021.07.020. Epub 2021 Aug 13. PMID 34393091
- See also: Genetic Modifiers of Cystic Fibrosis Lung and Liver Disease — http://cfmod.med.unc.edu/